CLINICAL TRIAL: NCT02966405
Title: The Establish of Trimester-specific Reference Ranges for Thyroid Tests in Pregnant Women and the Influence of Thyroid Disorders on Pregnancy and Its Outcomes.
Brief Title: The Establish of Specific Reference Ranges for Thyroid Tests in Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiaomei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Zhang, Director, Peking University International Hospital
Organization: Peking University International Hospital (Other)
Other Study IDs: PekingUIH
Record Dates: First submitted 2016-10-24; First posted 2016-11-17 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Diseases Pregnancy Thyroid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy pregnant women: A descriptive analysis involving 300 healthy pregnant women according NACB to the establish of trimester-specific reference ranges for thyroid tests in pregnant women.
- Normal pregnant population: According to the selection criteria, 700 cases were selected as the normal pregnant population to establish a self-sequential longitudinal reference range. The aim of this study to monitor the change of thyroid function and antibody during the course of pregnancy in those who suffer from various thyroid disorders and normal control.

SUMMARY:
A descriptive analysis involving 300 healthy pregnant women to the establish of trimester-specific reference ranges for thyroid tests in pregnant women. 700 cases were selected as the normal pregnant population to establish a self-sequential longitudinal reference range.

DETAILED DESCRIPTION:
A descriptive analysis involving 300 healthy pregnant women according NACB to the establish of trimester-specific reference ranges for thyroid tests in pregnant women. According to the selection criteria, 700 cases were selected as the normal pregnant population to establish a self-sequential longitudinal reference range. The aim of this study to monitor the change of thyroid function and antibody during the course of pregnancy in those who suffer from various thyroid disorders and normal control.

ELIGIBILITY:
Inclusion Criteria:

1. The people who lived in the city more than five years, aged between 19 and 45, or the single pregnancy women who registered or checked in Peking University international hospital would be enrolled.
2. The pregnancy confirmed by the ultrasound or blood HCG test.
3. In order to build a pregnancy reference range of normal pregnant women who must meet the NACB standard.

Exclusion Criteria:

1. The history of thyroid disorders.
2. Goiter.
3. Oral contraceptives or any drugs affected the function of thyroid.
4. With other chronic autoimmune disease, malignant tumor, blood disease, etc
5. Twin pregnancies and multiple pregnancies

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A descriptive analysis involving 300 healthy pregnant women according NACB to the establish of trimester-specific reference ranges for thyroid tests in pregnant women. According to the selection criteria, 700 cases were selected as the normal pregnant population to establish a self-sequential longitudinal reference range. The aim of this study to monitor the change of thyroid function and antibody during the course of pregnancy in those who suffer from various thyroid disorders and normal control.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Detection the FT3,FT4,TSH,TPOAb of the pregnant women in trimester of pregnancy. | up to 2 years
  Detection the FT3,FT4,TSH,TPOAb of the pregnant women in trimester of pregnancy.

SECONDARY OUTCOMES:
The influence of thyroid disorders on pregnancy. | up to 2 years
  Pregnant women:subclinical hypothyroidism,hypertension of pregnancy, eclampsia gravidarum, gestational diabetes mellitus, abortion, stillbirth.
The influence of thyroid disorders its outcomes. | up to 2 years
  Newborn:neonatal death,neonatal respiratory distress syndrome, low birth weight, macrosomia,et al.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao M zhang, Chief, Study Chair — Peking University International Hospital
Locations (2):
- China (2):
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Changping, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao D, Chai S, Yuan N, Sun J, Zhao X, Zhang X. Triglyceride-glycaemic index: Insights into predicting fetal macrosomia and its interaction with gestational diabetes mellitus: A cohort study of Chinese pregnant women. Eur J Clin Invest. 2024 Dec;54(12):e14300. doi: 10.1111/eci.14300. Epub 2024 Aug 13. PMID 39136403
- [Derived] Zhang X, Yuan N, Sun J, Zhao X, Du J, Nan M, Zhang Q, Ji L. Association Between Iodine Nutritional Status and Adverse Pregnancy Outcomes in Beijing, China: a Single-Center Cohort Study. Biol Trace Elem Res. 2022 Jun;200(6):2620-2628. doi: 10.1007/s12011-021-02887-9. Epub 2021 Sep 27. PMID 34570342
- [Derived] Yuan N, Sun J, Li Z, Chai S, Zhang X, Ji L. Relationship between anti-thyroid peroxidase antibody positivity and pregnancy-related and fetal outcomes in Euthyroid women: a single-center cohort study. BMC Pregnancy Childbirth. 2020 Aug 26;20(1):491. doi: 10.1186/s12884-020-03176-4. PMID 32847542